CLINICAL TRIAL: NCT03660514
Title: Jovenes Sanos: Preventing IPV and Reproductive Coercion Among Underserved Adolescents
Brief Title: Jovenes Sanos: Preventing IPV and RC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Comision de Salud Fronteriza Mexico - Estados Unidos (Unknown); Secretaria de Salud de Baja California (Unknown)
Responsible Party: Principal Investigator, Argentina Servin, MD, MPH, Assistant Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 161741; K23HD084756-01A1 (NIH)
Record Dates: First submitted 2018-08-28; First posted 2018-09-06 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Unintended Pregnancy; Family Planning; Intimate Partner Violence (IPV)
Keywords: Reproductive Coercion; Gender-based violence; Contraception; Clinic-based screening for IPV; Clinic-based counseling
MeSH Terms: interventions — cpsf4 protein, zebrafish

STUDY DESIGN:
Intervention Model Description: The Jovenes Sanos study will take place in two urban clinics in Tijuana, Mexico for all clients receiving voluntary FP counseling. The intervention study will involve a matched cluster control trial. Two clinics will serve as the intervention sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Family Planning (No Intervention): Counseling Clients receive standard FP counseling services.
- Jovenes Sanos Intervention in FP Counseling (Experimental): Clients receive the Jovenes Sanos intervention in addition to standard FP counseling services.
  Interventions: Behavioral: Jovenes Sanos

INTERVENTIONS:
Behavioral: Jovenes Sanos — FP counselors in intervention clinics will a) provide counseling and education regarding risk of partner detection of FP methods, and women's and girls' strategies to use FP methods to minimize partner detection risk integrated into standard FP counseling, b) make brief inquiries to allow clients the opportunity to disclose experiences of RC and IPC (i.e., screening), c) provide method-specific counseling based on this information and the method chosen by the client, d) provide supported linkage of IPV survivors to local IPV support services (i.e. warm referral), and e) distribute palm-sized educational materials on RC and IPV, as well as IPV services.
  Other Names: ARCHES
  Arms: Jovenes Sanos Intervention in FP Counseling

SUMMARY:
The primary purpose of this research is to conduct a small matched cluster control trial of an intervention designed to address reproductive coercion and unintended pregnancy (ARCHES - Addressing Reproductive Coercion within Healthcare Settings) adapted to the Mexican cultural and family planning healthcare context ( renamed Jovenes Sanos) in order to provide initial data regarding acceptability, feasibility and efficacy in this high need low-and-middle-income country.

DETAILED DESCRIPTION:
The project consortium will implement the ARCHES model across two community health centers in Tijuana, Baja California, Mexico. A 2-armed pilot study of ARCHES (adapted) will be conducted with 80 female FP clients (40 intervention, 40 control) ages 16-20 drawn from 2 comparable community health centers randomly assigned to either intervention or control (i.e. standard of care). Baseline data will be collected prior to routine FP service delivery, with a short exit survey conducted immediately following the clients' FP appointment (ARCHES or standard FP counseling will be provided during this visit). Follow-up data will be collected at 3-months post-intervention. Data at each time point will be collected via a 30-minute audio computer-assisted self-interview (ACASI) in Spanish. Data will also be collected to assess qualities of program implementation (i.e., process evaluation) to ensure implementation of the program as intended as well as unforeseen barriers to implementation. Creation of procedures for data collection, review of quality control data, and interpretation of findings will occur in collaboration with the entire mentoring/training committee. In-depth interviews (IDIs) with female adolescent FP clients ages 16-20 with a recent IPV/RC (n= 20), and focus groups (FGs) (n=2; 6-8 participants per group) with FP counselors in 2 comparable urban community health centers to identify perceptions of prevalence and impact of IPV and RC among adolescent clients and barriers to identifying IPV and RC. FGs with FP counselors from the participating community health centers will be conducted (n=2; 6-8 participants per group). FP counselors from these community health centers will be purposely selected to participate based on having provided FP services for at least 10 female adolescent clients in the past 6 months. At intervention sites, FP counselors will deliver the intervention integrated into standard-of-care practice; at control sites FP counselors will deliver solely standard-of-care services. Analyses specific to participants ages 16-20 will provide findings to guide consideration of ARCHES as an effective strategy to improve the reproductive health and reduce GBV among adolescents in this region.

ELIGIBILITY:
Inclusion Criteria: a) Client seeking voluntary FP services at community health centers; b)Aged 16-20 years; c) Biologically female; d) Willing to complete baseline, exit, and 3-month follow-up survey; e) Able to provide informed consent; f) Literate in Spanish; g) Screened positive for recent RC; h) Reside in Tijuana and have no plans to move in the next 12 months; i) Having no cognitive impairment that may interfere with their decisions to participate in the project (using Folstein Mini-Mental Exam); j) Not have participated in the IDIs (qualitative phase).

Ages: 16 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Biologically Female seeking family planning services
Enrollment: 124 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Recent RC | Change from prior 3 months (baseline) and 3-month follow-up
  RC consisted of two elements, pregnancy coercion and birth control sabotage. Pregnancy coercion was assessed using via 5 dichotomous items. Birth control sabotage was assessed via 5 dichotomous items measuring experiences of partner interference with contraception to promote pregnancy.

SECONDARY OUTCOMES:
Intimate Partner Violence (IPV) | Prior 3 months and prior 12 months
  Recent IPV is defined as violence in the past 3 months and Past IPV as violence in the past 12 months with participant's primary partner. a) Physical IPV: "pushed, pulled, slapped, held you down; punched you with fist or something that could hurt you; kicked or dragged you; tried to strangle or burn you; threatened you with a knife, gun, other weapon; attacked you with knife, gun, other weapon?" b) Sexual IPV: "used verbal threats to force you to have sex; physically forced you to have sex; or coerced you to perform other sexual acts when you did not want to?".
Contraception discontinuation | Prior 6 months and 12 months
  Items assessing discontinuation of use of method of contraception that participant reported using during prior 6 months or 12 months
Contraception self-efficacy | Baseline and 3-month follow-up
  Modified HIV risk reduction self-efficacy scale, which measures participants' reports of belief that she can enact certain contraceptive behaviors. This is a 4-item scale where each item has a 3-point measure from 0-2 with a score of 2 being very confident, 1 being somewhat confident, and 0 being not at all confident, for a total score range of 0-8.
Contraception delivery | Immediate post-intervention
  Report of receiving modern contraception method during clinic visit immediately preceding survey.
Biased and coercive FP provider practices | Immediate post-intervention
  Items to assess whether specified coercive or discriminatory behaviors were experienced from a FP provider during clinic visit immediately preceding survey.
Knowledge of IPV services | Present, assessed at baseline, 3-month follow-up
  Items assessing reported knowledge of listed local services for women and girls experiencing IPV
Utilization of IPV services among those reporting IPV | Prior 3 months and 6 months
  Items assessing whether participant called or visited a listed local service for women or girls experiencing IPV- only assessed for participants reporting history of IPV.

CONTACTS AND LOCATIONS:
Overall Officials: Argentina E Servin, MD, MPH, Principal Investigator — Division of Infectious Diseases and Global Public Health, University of California, San Diego
Locations (3):
- Division of Infectious Diseases and Global Public Health, University of California, San Diego, La Jolla, California, United States
- Mexico (2):
  - Centro de Salud Florido Morita, Tijuana, Estado de Baja California
  - Centro de Salud Fransisco Villa, Tijuana, Estado de Baja California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Uysal J, Stockman JK, Miller E, Rocha-Jimenez T, Rangel GM, Mercado AP, Servin AE. "At Least I Didn't Get Raped": A Qualitative Exploration of IPV and Reproductive Coercion among Adolescent Girls Seeking Family Planning in Mexico. J Interpers Violence. 2022 Apr;37(7-8):NP4740-NP4761. doi: 10.1177/0886260520959571. Epub 2020 Nov 12. PMID 33183147